CLINICAL TRIAL: NCT03271268
Title: The Role of CARdiovascular biOmarkers (NT-pro-BNP and CD146) in Predicting Lung Edema in Severely Burned Patients
Brief Title: Cardiovascular Biomarkers and Lung Edema in Severe Burns Patients
Acronym: CAROLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Principal Investigator, Sabri SOUSSI, MD, Saint-Louis Hospital, Paris, France
Other Study IDs: StLouisFrance
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Burns
Keywords: Vascular filling; Fluid overload; Biomarkers; Lung edema
MeSH Terms: conditions — Burns; Edema; Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum bank : 1 sample (5 ml of blood): on admission and from day 1 to day 7 of admission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Burn injury leads to hypovolemic then distributive shock. Fluid resuscitation remains the cornerstone of initial treatment of burn shock. However, fluid rescucitation can lead to fluid overload, which manifests most notably as lung edema.

The peptide NT-pro-BNP, a biomarker of cardiac congestion secreted by the myocardium, as well as plasma CD146, an endothelial factor involved in angiogenesis and a marker of vascular congestion, may help identifying patients with risk of pulmonary edema and hypoxia .

Our hypothesis is that these biomarkers may predict the occurence of pulmonary edema in severe burns patients.

ELIGIBILITY:
Inclusion Criteria:

* Intubated mechanically-ventilated patients within the first 24 hours of admission
* And/or patients with total body surface area (TBSA) burn-injured >20 %
* And/or patients with at least 10% full-thickness burns
* And/or receiving vasopressors within the first 24 hours of admission
* And monitored by a PiCCO system (PiCCO-2 Pulsion Medical Systems AG, Munich, Germany)

Exclusion Criteria:

* Admission delay to ICU > 24 hours post burn
* Age less than 18 years
* Pregnancy
* Chronic renal impairment with a baseline eGFR < 15 ml/min
* Patients with chemical or electrical burns
* Coexisting non-burn trauma
* Patients moribund on admission or dead within 72 h from admission
* Patients with do-not-resuscitate orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely ill burn patients admitted to a tertiary referral burn center
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2017-08-06 (Actual); Primary Completion 2019-02-06 (Estimated); Study Completion 2019-04-06 (Estimated)

PRIMARY OUTCOMES:
Lung edema | During the first 7 days of admission
  Extravascular lung water (EVLW) > 10 mL/Kg as measured by transpulmonary thermodilution (TPTD)

SECONDARY OUTCOMES:
Hypoxemia | During the first 7 days of admission for mechanically-ventilated patients
  PaO2/FiO2 ratio of <200
Hypercapnia | During the first 7 days of admission for mechanically-ventilated patients
  PaCO2> 45 mmHg
Corrected minute ventilation > 10L/min | During the first 7 days of admission for mechanically-ventilated patients
  Minute ventilation × partial [Paco2]/40) > 10L/min
Multiple organ dysfunction syndrome (MODS) | During the first 7 days of admission
  Sequential Organ Failure Assessment score (SOFA) ≥ 8
28-day mortality | 28 days
90-day mortality | 90 days
Length of stay in the ICU | until 90 days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sabri Soussi, MD, Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (1):
- Sabri SOUSSI, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Soluble CD146, a new endothelial biomarker of acutely decompensated heart failure — https://www.ncbi.nlm.nih.gov/pubmed/?term=Soluble+CD146%2C+a+new+endothelial+biomarker+of+acutely+decompensated+heart+failure
- See also: Natriuretic peptide type B in burn intensive care — https://www.ncbi.nlm.nih.gov/pubmed/23425748
- See also: Plasma Levels of Soluble CD146 Reflect the Severity of Pulmonary Congestion Better Than Brain Natriuretic Peptide in Acute Coronary Syndrome — https://www.ncbi.nlm.nih.gov/pubmed/?term=Plasma+Levels+of+Soluble+CD146+Reflect+the+Severity+of+Pulmonary+Congestion+Better+Than+Brain+Natriuretic+Peptide+in+Acute+Coronary+Syndrome